CLINICAL TRIAL: NCT05094908
Title: Randomized Clinical Trial to Evaluate the Safety and Therapeutic Response of Two ARNICA TINCTURE Treatment Regimes in the Topical Treatment of Uncomplicated Cutaneous Leishmaniasis in Colombia
Brief Title: Arnica Tincture Fot the Treatment of Cutaneous Leishmaniasis
Acronym: ARNICA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: INNOVATION CORPORATION FOR THE DEVELOPMENT OF PRODUCTS FOR TROPICAL DISEASES (CIDEPRO) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEC02_2021
Record Dates: First submitted 2021-09-28; First posted 2021-10-26 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Leishmaniasis, Cutaneous
Keywords: Leishmaniasis; Cutaneous; Arnica tincture
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — Arnicae flos extract; Solutions

STUDY DESIGN:
Intervention Model Description: This is an open, randomized, non-comparative, exploratory study with two arms. After the informed consent process and the verification of eligibility criteria, the volunteers will be randomly assigned to one of the interventions (30- or 45-day arnica tincture regimen) of the study.
  All individuals will have a telephone follow-up in the middle of the treatment, in addition, follow-up visits will be made at the end of the therapy, on day 45 post-treatment ± 5 days, on day 60 post-treatment ± 5 days (optional visit), on days 90 post-treatment ± 14 days and 180 days post-treatment-14 + 28 days to evaluate the therapeutic response. The participant will keep a record of the daily application (morning, afternoon and evening) of the study medication to document its application.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regime 1 (30 days) (Active Comparator): Regimen 1: arnica tincture applied 3 times a day for 30 days (group 1). For both regimens, the participant applies the tincture in the morning, afternoon and evening, that is, three times a day.
  Interventions: Drug: Arnica Tincture
- Regime 2 (45 days) (Active Comparator): Regimen 2 arnica tincture applied 3 times a day for 45 days (group 2). For both regimens, the participant applies the tincture in the morning, afternoon and evening, that is, three times a day.
  Interventions: Drug: Arnica Tincture

INTERVENTIONS:
Drug: Arnica Tincture — Arnika tincture is a topical plant-based preparation legally authorized in Colombia and in the countries of the European community, the product of this study is Arnika tinktur Gehrlicher (5249), manufactured by Gehrlicher Pharmazeutische Extrakte GmbH, Germany. According to the European Pharmacopoeia, the solution is a 70% hydroethanolic tincture prepared from the flowers of A. montana L, and composed at least 0.04% of sesquiterpene lactones. Arnica tincture will be applied topically by each participant on all lesions until day 30 or 45, depending on the regimen to be evaluated.
  Other Names: topical solution

SUMMARY:
Cutaneous Leishmaniasis (CL) is a parasitic disease caused by more than 20 different species of the protozoan parasite Leishmania. CL generally begins with a papule at the sand fly bite site, increasing to form a nodule that progresses to ulceration, or a scaly or wart-like plaque, over a period of 1 to 3 months.

The exact incidence of CL is not known. An estimated 1.2 million cases / year in approximately 100 countries around the world suffer from different forms of CL. In general, most lesions become ulcerated during the course of the disease. Among the different species of the parasite that cause LC, L. tropica from the Old World and L. braziliensis from the New World are considered the most important due to the severity of the disease they produce and because they are more difficult to cure with medications currently available.

Since 2010, the World Health Organization has insisted on the need to work on products that become alternatives for the treatment of CL, especially in products that serve topical application because with them, the probability of systemic toxicity is lower , increasing patient safety.

Among the options for topical treatment are natural products that have been, are, and will be extremely important as sources of medicinal agents. In addition to natural products that have found direct medicinal application as pharmaceutical entities, many others can serve as chemical models or templates for the design, synthesis and semi-synthesis of novel substances for the treatment of human diseases.

Arnica montana L. is a plant with anti-echemotic, healing, anti-inflammatory, analgesic and antineuralgic properties; It is included in the Colombian vademecum of medicinal plants. In previous studies it has been observed that the contact of the ulcerated skin with the product for up to 60 days does not generate toxic effects at the local level (application site) or at the systemic level, so it can be considered safe for use. To date there are no human studies with CL.

Therefore, it is intended to evaluate the safety and tolerability of Arnica tincture in individuals with uncomplicated CL, by measuring the occurrence and severity analysis of local and systemic adverse events.

DETAILED DESCRIPTION:
Arnica tincture is a topical preparation based on the plant legally authorized in the countries of the European community, and it is included in the vademecun of medicinal plants in Colombia. The research product is the commercial phytotherapeutic product ARNICA TINTURA Gehrlicher 100 mL manufactured by Gehrlicher Pharmazeutische Extrakte GmbH. (www. https://www.wer-zu-wem.de/firma/gehrlicher-extrakte.html). The product will be imported from Germany through the University of Munster (project co-investigator).

According to the European Pharmacopoeia, the solution is a 70% hydroethanolic tincture prepared from the flowers of Arnica montana L, and composed at least 0.04% of sesquiterpene lactones. Sesquiterpenic lactones (helenalin and 11-α-13 dihydrohelenaline) are the constituents responsible for its anti-inflammatory activity, these molecules decrease inflammation mediated by the transcription factor NF-kB. There are other properties demonstrated in the literature such as antioxidant, antimicrobial or insecticidal activities.

Given the plant's anti-inflammatory, healing, anti-echemotic, analgesic and antineuralgic properties, in a previous study the leishmanicidal activity of arnica tincture was evaluated in vitro for intracellular amastigotes of L. braziliensis and L. tropica. Arnica tincture at a concentration of 4.8 mg / mL produced a decrease in the parasite load (amount of intracellular amastigotes) of 91.9% and 99.6% in cells infected by L. braziliensis and L. tropica, respectively. . The mean maximum Effective Concentrations (EC50) were determined at 2.9 ± 0.13 and 2.7 ± 0.02 respectively, and with selectivity indices> 69 and> 74, for L. braziliensis and L. tropica, respectively. This activity was validated in in vivo studies in hamsters experimentally infected with L. braziliensis. Applying the tincture once a day for 30 days produced a cure of 60 and for the remaining 40% of the hamsters a reduction of more than 80% of the lesions was observed (Robledo et al., 2018). When applied once a day for 60 days, 75% of the hamsters were cured and the remaining 25% showed improvements between 70 and 96% regarding the size of the lesion before treatment. According to the observations made, it is part of the natural evolution of the healing process that, during the first weeks of use of the compound and until the end of the treatment, a flattening of the edges is perceived, with intensification of the erythema, which produces a Optical sensation of enlargement of the lesion, which subsequently (from day 28) gives rise to the re-epithelialization process, which is slightly slower compared to traditional systemic schemes. The percentage of epithelialization of the lesion (s) is calculated by comparing the size of the ulcer at baseline against the size observed at the follow-up visit.

Arnica tincture is not cytotoxic on epithelial cells (Detroit) at any concentrations tested. In liver cells (HepG2) the tincture showed a slight cytotoxicity when evaluated at 100%, with a toxicity percentage of 75%. Weight, clinical appearance, and behavior data, as well as ALT, alkaline phosphatase, creatinine, and urea test results; and the histological studies obtained from the tests in hamsters allowed to conclude that the contact of the ulcerated skin with the product for up to 60 days does not generate toxic effects at the local level (application site) or at the systemic level, so it can be considered as safe for use. Corrosion and irritation tests to evaluate arnica skin tincture according to OECD guidelines suggest that it is neither corrosive nor irritating.

Although it is difficult to calculate accurately, it has been estimated that approximately 2 drops (80uL) of the solution will be used per cm2 in each application. If we consider an average lesion size of 4 cm2, a maximum of 320 uL is used X 3 times a day X 45 or 30 days = 43,200 uL or 28,800uL (equivalent to 43.2 or 28.8 mL) per lesion.

1. Main Objectives

   * Evaluate the safety and tolerability of Arnica tincture in individuals with uncomplicated CL, by measuring the occurrence and severity analysis of local and systemic ADs.
   * Evaluate the therapeutic response of Arnica tincture in individuals with uncomplicated CL, according to the percentage of individuals with initial clinical cure on day 90.

   Regimen 1: Arnica tincture applied 3 times a day for 30 days (Group 1: 4 weeks) Regimen 2: Arnica tincture applied 3 times a day for 45 days (Group 2: 6 weeks)
2. Secondary Objectives

   * Evaluate the frequency and severity of AEs associated with the use of the Arnica tincture solution.
   * Assess the status of the lesions over time, up to 100% epithelialization of ulcerated lesions and proportion of individuals with 100% epithelialization of non-ulcerated lesions over time.
   * Assess the relapse rate.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, of legal age, between 18 and 65 years old.
* With a confirmed parasitological diagnosis of CL in at least one lesion, performed at least through the following methods: 1) microscopic identification of amastigotes in the lesion tissue; 2) diagnosis of leishmania through PCR; 3) positive culture for promastigotes.
* Subjects with an injury that meets the following criteria:

  * Ulcer or nodule with a maximum size of 4 cm (the largest diameter).
  * Not located in the ear, face, near mucous membranes, joints, or in places where, in the opinion of the IP, the administration of the product is difficult to apply topically.
* Subjects with a maximum of 4 LC lesions.
* Injury with an evolution of less than 4 months according to the subject's history.
* Subjects who have given their CI in writing.
* At the discretion of the IP, the subject is able to understand and comply with the requirements of the study.
* Subjects who can attend control visits.

Exclusion Criteria:

* Women with a positive pregnancy test during the screening process, or breastfeeding, or women of childbearing potential who do not accept the use of contraceptives during treatment and up to 45 days after treatment.
* History of clinically significant medical problems or treatments that may interact negatively or positively with topical treatment for Leishmaniasis, including any immunocompromising conditions.
* Within 8 weeks (56 days) of starting the study treatment, having received treatment for Leishmaniasis with any type of medication, including Glucantime that probably, in the opinion of the PI, could modify the course of infection with Leishmania.
* Based on physical examinations performed, a diagnosis of CML has been or is suspected.
* Known or suspected history of hypersensitivity or idiosyncratic reactions to study treatment.
* Present the following laboratory alterations:

  * Serum creatinine above normal levels
  * ALT / AST levels 3 times above the normal value (according to the levels reported by the local laboratory).
* Subjects who do not want to keep study appointments or who cannot keep follow-up visits for up to six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-11-02 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Initial post-treatment healing | day 90
  defined as 100% epithelialization of the lesion (s) by day 90 post-treatment.

SECONDARY OUTCOMES:
Number of participants with Final post-treatment Healing | day 180
  initial healing without relapse and / or mucosal compromise at the 180th day post-treatment evaluation
Number of participants with lesions that relapse | day 180
  lesion that achieves 100% epithelialization by Day 90 post-treatment and then returned to show activity by day 180 post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan D Velez, PhD, Principal Investigator — Director PECET
Locations (1):
- Program for Research and Control in Tropical Diseases - PECET, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robledo SM, Velez ID, Schmidt TJ. Arnica Tincture Cures Cutaneous Leishmaniasis in Golden Hamsters. Molecules. 2018 Jan 12;23(1):150. doi: 10.3390/molecules23010150. PMID 29329207
- [Background] Guidelines of the International Conference on Harmonization - Good Clinical Practice: Consolidated Guide (ICH E6), E6(R2) Current Step 4 version dated 9 November 2016
- [Background] Management of Safety Information from Clinical Trials Report of CIOMS Working Group VI, Geneva 2005, Organizations of Medical Sciences (CIOMS) ISBN 92 9036 079 8
- [Background] Blum J, Lockwood DN, Visser L, Harms G, Bailey MS, Caumes E, Clerinx J, van Thiel PP, Morizot G, Hatz C, Buffet P. Local or systemic treatment for New World cutaneous leishmaniasis? Re-evaluating the evidence for the risk of mucosal leishmaniasis. Int Health. 2012 Sep;4(3):153-63. doi: 10.1016/j.inhe.2012.06.004. PMID 24029394
- [Background] Blum J, Desjeux P, Schwartz E, Beck B, Hatz C. Treatment of cutaneous leishmaniasis among travellers. J Antimicrob Chemother. 2004 Feb;53(2):158-66. doi: 10.1093/jac/dkh058. Epub 2004 Jan 16. PMID 14729756
- [Background] Soto J, Rea J, Balderrama M, Toledo J, Soto P, Valda L, Berman JD. Efficacy of miltefosine for Bolivian cutaneous leishmaniasis. Am J Trop Med Hyg. 2008 Feb;78(2):210-1. PMID 18256415
- [Background] WHO technical report series; no. 949. Control of the leishmaniasis: report of a meeting of the WHO Expert Committee on the Control of Leishmaniases, Geneva, 22-26 March 2010
- [Background] Silva NS, Muniz VD. [Epidemiology of American tegumentary leishmaniasis in the State of Acre, Brazilian Amazon]. Cad Saude Publica. 2009 Jun;25(6):1325-36. doi: 10.1590/s0102-311x2009000600015. Portuguese. PMID 19503963
- [Background] Almeida OL, Santos JB. Advances in the treatment of cutaneous leishmaniasis in the new world in the last ten years: a systematic literature review. An Bras Dermatol. 2011 May-Jun;86(3):497-506. doi: 10.1590/s0365-05962011000300012. English, Portuguese. PMID 21738967
- [Background] Tiuman TS, Santos AO, Ueda-Nakamura T, Filho BP, Nakamura CV. Recent advances in leishmaniasis treatment. Int J Infect Dis. 2011 Aug;15(8):e525-32. doi: 10.1016/j.ijid.2011.03.021. Epub 2011 May 24. PMID 21605997
- [Background] Herwaldt BL. Leishmaniasis. Lancet. 1999 Oct 2;354(9185):1191-9. doi: 10.1016/S0140-6736(98)10178-2. PMID 10513726
- [Background] Velez I, Lopez L, Sanchez X, Mestra L, Rojas C, Rodriguez E. Efficacy of miltefosine for the treatment of American cutaneous leishmaniasis. Am J Trop Med Hyg. 2010 Aug;83(2):351-6. doi: 10.4269/ajtmh.2010.10-0060. PMID 20682881
- [Background] Croft SL, Seifert K, Yardley V. Current scenario of drug development for leishmaniasis. Indian J Med Res. 2006 Mar;123(3):399-410. PMID 16778319
- [Background] Pearson, R. D., A. De Queiroz Sousa, and S. M. B. Jeronimo. 2001. Leishmania species: visceral (kala-azar), cutaneous and mucosal leishmaniasis, p. 2831-2845. In G. L. Mandell, J. E. Bennett, and R. Dolin (ed.), Principles and practice of infectious diseases. Churchill Livingstone, New York, N.Y
- [Background] Votypka J, Kasap OE, Volf P, Kodym P, Alten B. Risk factors for cutaneous leishmaniasis in Cukurova region, Turkey. Trans R Soc Trop Med Hyg. 2012 Mar;106(3):186-90. doi: 10.1016/j.trstmh.2011.12.004. Epub 2012 Jan 26. PMID 22284721
- [Background] Alvar J, Velez ID, Bern C, Herrero M, Desjeux P, Cano J, Jannin J, den Boer M; WHO Leishmaniasis Control Team. Leishmaniasis worldwide and global estimates of its incidence. PLoS One. 2012;7(5):e35671. doi: 10.1371/journal.pone.0035671. Epub 2012 May 31. PMID 22693548
- [Background] Reveiz L, Maia-Elkhoury AN, Nicholls RS, Romero GA, Yadon ZE. Interventions for American cutaneous and mucocutaneous leishmaniasis: a systematic review update. PLoS One. 2013 Apr 29;8(4):e61843. doi: 10.1371/journal.pone.0061843. Print 2013. PMID 23637917
- [Background] Lee SA, Hasbun R. Therapy of cutaneous leishmaniasis. Int J Infect Dis. 2003 Jun;7(2):86-93. doi: 10.1016/s1201-9712(03)90002-6. PMID 12839708
- [Background] Lopez L, Robayo M, Vargas M, Velez ID. Thermotherapy. An alternative for the treatment of American cutaneous leishmaniasis. Trials. 2012 May 17;13:58. doi: 10.1186/1745-6215-13-58. PMID 22594858
- [Background] Velasco-Castrejon O, Walton BC, Rivas-Sanchez B, Garcia MF, Lazaro GJ, Hobart O, Roldan S, Floriani-Verdugo J, Munguia-Saldana A, Berzaluce R. Treatment of cutaneous leishmaniasis with localized current field (radio frequency) in Tabasco, Mexico. Am J Trop Med Hyg. 1997 Sep;57(3):309-12. doi: 10.4269/ajtmh.1997.57.309. PMID 9311641
- [Background] Wagner S, Suter A, Merfort I. Skin penetration studies of Arnica preparations and of their sesquiterpene lactones. Planta Med. 2004 Oct;70(10):897-903. doi: 10.1055/s-2004-832613. PMID 15490315
- [Background] Assessment report on Arnica montana L., ﬂos, European Medicines Agency (Science medicines agency), 9 July 2013 EMA/HMPC/198794/2012 Committee on Herbal Medicinal Products (HMPC)
- [Background] Iannitti T, Morales-Medina JC, Bellavite P, Rottigni V, Palmieri B. Effectiveness and Safety of Arnica montana in Post-Surgical Setting, Pain and Inflammation. Am J Ther. 2016 Jan-Feb;23(1):e184-97. doi: 10.1097/MJT.0000000000000036. PMID 25171757
- [Derived] Robledo SM, Lopez L, Quintero J, Tabares Y, Garces AC, Rios-Echavarria S, Soto E, Velez ID, Schmidt TJ. A phase Ib/II clinical study to evaluate the safety and efficacy of topical Arnica tincture to treat non-complicated cutaneous leishmaniasis in Colombia. PLoS Negl Trop Dis. 2025 Aug 18;19(8):e0013123. doi: 10.1371/journal.pntd.0013123. eCollection 2025 Aug. PMID 40825042
- See also: Ministry of Social Protection, 2008. Colombian Vademecum of Medicinal Plants — https://www.minsalud.gov.co/sites/rid/Lists/BibliotecaDigital/RIDE/VS/PP/SA/vademecum-colombiano-plantas-medicinales.pdf
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — http://ctep.cancer.gov
- See also: Pan American Health Organization, PAHO. Leishmaniasis in the Americas: Recommendations for treatment. 2013 — http://www.paho.org/hq/index.php?option=com_docman&task=doc_view&gid=22226&Itemid